CLINICAL TRIAL: NCT06554678
Title: THRIVE Improves Early Postoperative Atelectasis in Long-Time Non-Tracheal Intubation Anesthesia for Gastrointestinal Endoscopy: a Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Ju Gao, Study Director, Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024ky033
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-10

CONDITIONS: Early Postoperative Atelectasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transnasal humidified rapid insufflation ventilatory exchange（THRIVE） group (Experimental)
  Interventions: Procedure: Transnasal humidified rapid insufflation ventilatory exchange（THRIVE）
- conventional oxygen mask group (Active Comparator)
  Interventions: Procedure: conventional oxygen mask

INTERVENTIONS:
Procedure: Transnasal humidified rapid insufflation ventilatory exchange（THRIVE） — Transnasal humidified rapid insufflation ventilatory exchange（THRIVE）
  Arms: Transnasal humidified rapid insufflation ventilatory exchange（THRIVE） group
Procedure: conventional oxygen mask — conventional oxygen mask
  Arms: conventional oxygen mask group

SUMMARY:
This study aims to explore the clinical effect of THRIVE in improving early postoperative atelectasis in patients undergoing long-term non-intubated anesthesia gastrointestinal endoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Multiple polyps resection, ESD(Endoscopic Submucosal Dissection) , EMR(Endoscopic Mucosal Resection), enteroscopy and other gastrointestinal endoscopic diagnosis and treatment were performed
2. The duration of anesthesia is more than 30 minutes, that is, from induction to withdrawal of anesthesia
3. ASA(American Society of Anesthesiologists) ≤ II 4.18kg/m2<BMI<30 kg/m2

5.Informed consent, voluntary participation in the experiment, and signed by the subject informed consent

Exclusion Criteria:

1. ASA classification ≥ III;
2. History of previous lung or nasal surgery;
3. History of chronic obstructive pulmonary disease (COPD) or restrictive lung disease;
4. History of obstructive sleep apnea syndrome;
5. History of upper airway obstruction;
6. History of head and neck radiation therapy;
7. Significant nasal septum deviation;
8. Active infection (defined as a white blood cell count >10*10^9 or a body temperature >38°C);
9. Gastrointestinal perforation;
10. Combined use of other anesthetic methods or inhalation anesthetics outside of non-intubated intravenous anesthesia;
11. Concurrent other medical procedures besides the prescribed gastrointestinal endoscopic procedures, such as ERCP(Endoscopic Retrograde Cholangiopancreatography);
12. Severe communication disorders due to conditions like severe hearing impairment or dementia;
13. Disagreement with participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-18 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of atelectasis | Early postoperative period
  Lung ultrasound examination was performed before anesthesia induction (T1) and immediately after surgery (T2), and patients' modified lung ultrasound score (LUSS) was recorded.

SECONDARY OUTCOMES:
Diaphragm movement | Before anesthesia induction (T1) and immediately after surgery (T2)
Heart rate (HR) | Baseline，during surgery and arrived at PACU
  Throughout the procedure, the heart rate (HR) was continuously monitored.
Pulse oxygen saturation (SpO2) | Baseline，during surgery and arrived at PACU
  Throughout the procedure, the pulse oxygen saturation (SpO2) were continuously monitored.
Mean blood pressure (MBP) | Baseline，during surgery and arrived at PACU
  Throughout the procedure, the mean blood pressure (MBP) was measured at 3-minute intervals.
Patient satisfaction levels | After the patient is awake
  The patients express their satisfaction with procedures on a numerical rating scale, ranging from 0 to 10, where 0 is the minimum and 10 is the maximum satisfaction level.
Endoscopist satisfaction levels | After the surgery
  The Endoscopists express their satisfaction with procedures on a numerical rating scale, ranging from 0 to 10, where 0 is the minimum and 10 is the maximum satisfaction level.
Adverse Events (AEs) During Surgery and PACU | During surgery and PACU
  radycardia; Hypertension; Hypotension; Hypoxemia; Aspiration and Regurgitation
Adverse Events (AEs) Within 7 Days Post-Operatively | Within 7 days after surgery
  Fever; Cough and Sputum Production; Antibiotic Usage
PACU Stay Duration | The time from entering PACU to improving Aldrete score ≥9
Length of Hospital Stay | The time from admission to discharge
Dosage of propofol | During surgery
Dosage of remifentanil | During surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China